CLINICAL TRIAL: NCT01794793
Title: An Open Label, Multi-center Pasireotide Roll-over Protocol for Patients Who Have Completed a Previous Novartis-sponsored Pasireotide Study and Are Judged by the Investigator to Benefit From Continued Pasireotide Treatment
Brief Title: Study to Allow Access to Pasireotide for Patients Benefiting From Pasireotide Treatment in Novartis-sponsored Studies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230B2412
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Results first posted 2024-08-28 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Cushing's Disease; Acromegaly; Neuroendocrine Tumors; Pituitary Tumors; Ectopic ACTH Secreting (EAS) Tumors; Dumping Syndrome; Prostate Cancer; Melanoma Negative for bRAF; Melanoma Negative for nRAS
Keywords: SOM230,; roll-over study; pasireotide LAR; Cushing's disease; Acromegaly; neuroendocrine tumorsNETs; pituitary tumors; Ectopic ACTH secreting; EAS; Dumping Syndrome; metastatic prostate cancer, metastatic melanoma; bRAF; nRAS
MeSH Terms: conditions — Pituitary ACTH Hypersecretion; Acromegaly; Neuroendocrine Tumors; Pituitary Neoplasms; Neoplasms; Dumping Syndrome; Prostatic Neoplasms; Melanoma | interventions — pasireotide; Cabergoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pasireotide subcutaneous (Experimental): 0.3mg, 0.6mg and 0.9mg. Doses to be taken BID or TID, dependent on parent study guidelines. Cabergoline may be combined in this arm for Cushing's Disease and Acromegaly patients.
  Interventions: Drug: Pasireotide; Drug: Cabergoline
- Pasireotide Long Acting Release (LAR) (Experimental): 10mg, 20mg, 40mg and 60mg. All doses to be taken q28days. Strength is dependent on parent study guidelines.
  Interventions: Drug: Pasireotide LAR

INTERVENTIONS:
Drug: Pasireotide — Administered subcutaneously in strengths 0.3mg, 0.6mg and 0.9mg. Doses to be taken BID or TID, dependent on parent study guidelines.
  Other Names: SOM230; Signifor
  Arms: Pasireotide subcutaneous
Drug: Cabergoline — Cabergoline tablet 0.5mg or 1.0mg taken by mouth once daily may be combined with subcutaneous formulation of pasireotide for Cushing's Disease or Acromegaly. Dose is dependent on parent study guidelines.
  Other Names: dostinex
  Arms: Pasireotide subcutaneous
Drug: Pasireotide LAR — Long Acting Release is administered by a single intramuscular (i.m.) monthly injection. The strengths are 10mg, 20mg, 40mg and 60mg. All doses to be taken q28days. Strength is dependent on parent study guidelines.
  Other Names: SOM230; Signifor
  Arms: Pasireotide Long Acting Release (LAR)

SUMMARY:
The purpose of this study is to allow continued use of pasireotide in patients who are on pasireotide treatment in a Novartis-sponsored study and are benefiting from the treatment as judged by the investigator.

DETAILED DESCRIPTION:
This is a multi-center, open label, phase IV study to provide continued supply of pasireotide to patients being treated in a current Novartis-sponsored study and who are benefiting from treatment with pasireotide alone or in combination with another treatment for Cushing's Disease and Acromegaly . Eligible patients are to be consented and can then continue treatment with pasireotide alone or in combination with another treatment for Cushing's Disease and Acromegaly in this protocol. All patients at their scheduled visits will have drug dispensing information and reported adverse events and serious adverse events collected.

A patient will reach the end of study when pasireotide treatment is permanently discontinued and the end of treatment visit has been performed. All patients must be followed up for safety evaluations for 3 months following the last dose of pasireotide LAR treatment and for 1 month following the last dose of pasireotide s.c. treatment.

The study is expected to remain open for approximately 10 years or until such time that enrolled patients no longer need treatment with pasireotide or are able to obtain commercial supply according to local regulations for their medical condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is currently participating in a Novartis-sponsored study receiving pasireotide (LAR and/or s.c.) on monotherapy or combination therapy (for Cushing's Disease or Acromegaly), and has fulfilled all required assessments in the parent study and patients that are benefiting from the study treatment have no other alternatives.
2. Patient is currently benefiting from the treatment with pasireotide, as determined by the investigator
3. Patient has demonstrated compliance, as assessed by the investigator, with the parent study requirements.
4. Willingness and ability to comply with scheduled visits, treatment plans and any other study procedures.
5. Written informed consent obtained prior to enrolling in roll-over study and receiving study medication.

   * If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.

Exclusion Criteria:

1. Patient has been permanently discontinued from pasireotide study treatment in the parent study due to unacceptable toxicity, non-compliance to study procedures, withdrawal of consent or any other reason.
2. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
3. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during the study treatment and for 30 days after the final dose of pasireotide s.c. and 84 days after the final dose of pasireotide LAR. Highly effective contraception is defined as either:

   * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
   * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
   * Male sterilization (at least 6 months prior to enrolling). For female patients on the study the vasectomized male partner should be the sole partner for that patient.
   * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
   * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
   * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.
   * Sexually active males, unless they use a condom during intercourse while taking drug and for 1 months after pasireotide s.c. last dose and 3 months after pasireotide LAR last dose, should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2013-06-10 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Recordati, Study Director — Recordati AG
Locations (89):
- United States (7):
  - Ximed Research SC - SOM230B2412, La Jolla, California
  - Cedars Sinai Medical Center Cedars Sinai 4, Los Angeles, California
  - Stanford Universtiy Medical Center Stanford Hospital & Clinics, Stanford, California
  - University of Michigan Comprehensive Cancer Center SC-2, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center SC, New York, New York
  - Virginia Endocrinology Research SC, Chesapeake, Virginia
  - Swedish Cancer Institute Swedish Cancer Institute (SC), Seattle, Washington
- Argentina (2):
  - Recordati Investigative Site, CABA, Buenos Aires
  - Recordati Investigative Site, Mar del Plata, Buenos Aires
- Belgium (7):
  - Recordati Investigative Site, Edegem, Antwerpen
  - Recordati Investigative Site, Bruges
  - Recordati Investigative Site, Brussels
  - Recordati Investigative Site, Ghent
  - Recordati Investigative Site, Leuven
  - Recordati Investigative Site, Liège
  - Recordati Investigative Site, Wilrijk
- Brazil (7):
  - Recordati Investigative Site, Fortaleza, Ceará
  - Recordati Investigative Site, Curitiba, Paraná
  - Recordati Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Recordati Investigative Site, Porto Alegre, Rio Grande do Sul
  - Recordati Investigative Site, Joinville, Santa Catarina
  - Recordati Investigative Site, Botucatu, São Paulo
  - Recordati Investigative Site, São Paulo, São Paulo
- Recordati Investigative Site, Sofia, Bulgaria
- Canada (3):
  - Recordati Investigative Site, Halifax, Nova Scotia
  - Recordati Investigative Site, London, Ontario
  - Recordati Investigative Site, Montreal, Quebec
- France (8):
  - Recordati Investigative Site, Toulouse, Cedex 9
  - Recordati Investigative Site, Angers
  - Recordati Investigative Site, Bron
  - Recordati Investigative Site, Le Kremlin-Bicêtre
  - Recordati Investigative Site, Lille
  - Recordati Investigative Site, Marseille
  - Recordati Investigative Site, Pessac
  - Recordati Investigative Site, Pierre-Bénite
- Germany (6):
  - Recordati Investigative Site, Berlin
  - Recordati Investigative Site, Hamburg
  - Recordati Investigative Site, München
  - Recordati Investigative Site, Tübingen
  - Recordati Investigative Site, Ulm
  - Recordati Investigative Site, Würzburg
- Recordati Investigative Site, Athens, GR, Greece
- Recordati Investigative Site, Budapest, Hungary
- India (2):
  - Recordati Investigative Site, Bangalore, Karnataka
  - Recordati Investigative Site, Vellore, Tamil Nadu
- Recordati Investigative Site, Petah Tikva, Israel
- Italy (5):
  - Recordati Investigative Site, Ancona, AN
  - Recordati Investigative Site, Genova, GE
  - Milano Investigative Site, Milan, MI
  - Recordati Investigative Site, Padua, PD
  - Recordati Investigative Site, Roma, RM
- Japan (6):
  - Recordati Investigative Site, Nagoya, Aichi-ken
  - Recordati Investigative Site, Maebashi, Gunma
  - Recordati Investigative Site, Kobe, Hyōgo
  - Recordati Investigative Site, Nankoku, Kochi
  - Recordati Investigative Site, Kyoto, Kyoto
  - Recordati Investigative Site, Suita, Osaka
- Malaysia (2):
  - Recordati Investigative Site, Kuala Lumpur
  - Recordati Investigative Site, Pulau Pinang
- Mexico (4):
  - Recordati Investigative Site, Guadalajara, Jalisco
  - Recordati Investigative Site, Mexico City, Mexico City
  - Recordati Investigative Site, Durango
  - Recordati Investigative Site, Mexico City
- Recordati Investigative Site, Groningen, Netherlands
- Recordati Investigative Site, San Isidro, Lima region, Peru
- Poland (4):
  - Recordati Investigative Site, Gdansk
  - Recordati Investigative Site, Poznan
  - Recordati Investigative Site, Warsaw
  - Recordati Investigative Site, Wroclaw
- Recordati Investigative Site, Porto, Portugal
- Recordati Investigative Site, Bucharest, Romania
- Russia (4):
  - Recordati Investigative Site, Barnaul
  - Recordati Investigative Site, Moscow
  - Recordati Investigative Site, Saint Petersburg
  - Recordati Investigative Site, Tyumen
- Recordati Investigative Site, Seoul, South Korea
- Spain (2):
  - Recordati Investigative Site, Alicante, Valencia
  - Recordati Investigative Site, Barcelona
- Switzerland (2):
  - Recordati Investigative Site, Lausanne
  - Recordati Investigative Site, Zurich
- Recordati Investigative Site, Taichung, Taiwan
- Thailand (2):
  - Recordati Investigative Site, Bangkok
  - Recordati Investigative Site, Songkhla
- Turkey (Türkiye) (6):
  - Recordati Investigative Site, Istanbul, TUR
  - Recordati Investigative Site, Ankara
  - Recordati Investigative Site, Antalya
  - Recordati Investigative Site, Istanbul
  - Recordati Investigative Site, Izmir
  - Recordati Investigative Site, Kocaeli

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No target number of patients pre-specified for this study
Groups:
- All Subjects: Patients who were treated with and had benefitted from pasireotide in the parent studies remained enrolled in this study and were elegible for the analysis
Period: Treatment Period
Arm/Group | All Subjects
Started | 337
Completed | 239
Not Completed | 98
Not completed — Withdrawal by Subject | 24
Not completed — Lack of Efficacy | 22
Not completed — Adverse Event | 17
Not completed — Physician Decision | 14
Not completed — Lost to Follow-up | 7
Not completed — Death | 6
Not completed — Protocol Violation | 5
Not completed — administrative problem | 3
Period: Post-treatment Follow-up
Arm/Group | All Subjects
Started | 149 (188/ 337 patients did not enter the post-treatment follow-up safety evaluation)
Completed | 110
Not Completed | 39
Not completed — Lack of Efficacy | 14
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 6
Not completed — administrative problem | 5
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 337
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 305
  >=65 years | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190
  Male | 147
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events to Evaluate Long Term Safety Data
Description: Collect long term safety data, i.e. SAEs and AEs. SAES will be reviewed and reported as part of the regular pharmacovigilance activities.
Time Frame: Baseline up to approximately 10 years
Population: The Safety Set included all patients who received at least one dose of study medication (pasireotide) after enrolling into the roll-over protocol
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 337
participants
  AEs : All grades | 265
  AEs : Grades ≥3 | 102
  Treatment-related AEs : All grades | 127
  Treatment-related AEs : Grades ≥3 | 39
  SAEs : All grades | 91
  SAEs : Grades ≥3 | 72
  Fatal SAEs : All grades | 8
  Fatal SAEs : Grades ≥3 | 8
  Treatment-related fatal SAEs : All grades | 0
  Treatment-related fatal SAEs : Grades ≥3 | 0
  AEs leading to discontinuation : All grades | 20
  AEs leading to discontinuation : Grades ≥3 | 11
  Treatment-related AEs leading to discontinuation : All grades | 16
  Treatment-related AEs leading to discontinuation : Grades ≥3 | 7
  AEs leading to dose adjustment/interruption : All grades | 39
  AEs leading to dose adjustment/interruption : Grades ≥3 | 13
  AEs requiring additional therapy : All grades | 220
  AEs requiring additional therapy : Grades ≥3 | 62

2. Secondary Outcome: Percentage of Patients With Clinical Benefit as Assessed by the Investigator
Description: Efficacy was assessed by the investigator at each scheduled visit using a binary (yes/no) response confirming the investigator's judgement of clinical benefit (via the question: "Does investigator confirm that the subject continues to have clinical benefit from the study treatment"). No other measures of efficacy were used in this study.
Time Frame: Baseline up to approximately 10 years
Population: Number of patients judged by the investigator to be clinically benefitting from treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Pasireotide Long Acting Release (LAR): 10mg, 20mg, 40mg and 60mg. All doses to be taken q28days i.m. Strength is dependent on parent study guidelines
Arm/Group | Pasireotide Subcutaneous | Pasireotide Long Acting Release (LAR)
Number analyzed (Participants) | 38 | 299
Participants
  Month 3 | 29 | 256
  Month 6 | 28 | 250
  Month 12 | 21 | 234
  Month 18 | 19 | 216
  Month 24 | 17 | 198
  Month 36 | 14 | 177
  Month 48 | 15 | 162
  Month 60 | 12 | 140
  Month 72 | 12 | 98
  Month 84 | 8 | 21
  Month 96 | 5 | 1
  Month 108 | 5 | 1
  Month 120 | 2 | 0

ADVERSE EVENTS:
Time Frame: Pasireotide s.c.: From start of study treatment up to 1 month after study treatment discontinuation (about 10 years) Pasireotide LAR: From start of study treatment up to 3 months after study treatment discontinuation (about 10 years)
Description: Safety was monitored by collecting AEs/SAEs at every visit and throughout the study period (not limited to patient contact times) according to the sponsor's routine safety monitoring practices. Patients might have safety assessments performed by the clinic's local laboratory as per investigators judgement and standard of care at any time during the study period.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 8/337
Serious Adverse Events (participants affected / at risk) | 91/337
Other Adverse Events (participants affected / at risk) | 220/337
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=337)
Cholelithiasis (Hepatobiliary disorders) | 9
Cholecystitis (Hepatobiliary disorders) | 5
COVID-19 (Infections and infestations) | 8
Cellulitis (Infections and infestations) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Cardiorespiratory arrest (Cardiac disorders) | 1
Myocardial Ischaemia (Cardiac disorders) | 1
Syringomyelia (Congenital, familial and genetic disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hyperadrenocorticism (Endocrine disorders) | 1
Cataract (Eye disorders) | 1
Abdominal adhesion (Gastrointestinal disorders) | 1
Abdominal fat apron (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Large Intestin Polyp (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stasis Syndrome (Gastrointestinal disorders) | 1
Umbelical hernia (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
General physical health deterioration (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 1
Cholangitis chronic (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Hydrocholecystitis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 3
COVID-19 pneumonia (Infections and infestations) | 2
Septic shock (Infections and infestations) | 2
Abscess jaw (Infections and infestations) | 1
Acute sinusitis (Infections and infestations) | 1
Coronavirus infection (Infections and infestations) | 1
Diarrhoea infectious (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Infected dermal cyst (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneunomia pseudomonal (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Suspected COVID-19 (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Meniscus injury (Infections and infestations) | 1
Poisoning (Injury, poisoning and procedural complications) | 1
Suture related complication (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Hepatic enzyme increased (Investigations) | 1
Weight decreased (Infections and infestations) | 1
Diabetic ketoacidosis (Infections and infestations) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Diabetic ketosis (Metabolism and nutrition disorders) | 1
Diabetic metabolic decompesation (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pituitary tumour recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Epilepsy (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Dementia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Hypoglycaemic coma (Nervous system disorders) | 1
Hypoglycaemic seizure (Nervous system disorders) | 1
Myasthenia gravis (Nervous system disorders) | 1
Transient Ischaemic attack (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Mental fatigue (Psychiatric disorders) | 1
Psychiatric decompensation (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Distributive shock (Vascular disorders) | 1
Hypertensive emergency (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral embolism (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=337)
Nasopharyngitis (Infections and infestations) | 32
Back pain (Musculoskeletal and connective tissue disorders) | 30
Hypertension (Vascular disorders) | 25
Hyperglycaemia (Metabolism and nutrition disorders) | 23
Headache (Nervous system disorders) | 22
Covid-19 (Infections and infestations) | 20
Urinary tract infection (Infections and infestations) | 19
Influenza (Infections and infestations) | 18
Diabetes mellitus (Metabolism and nutrition disorders) | 18
Diarrhoea (Gastrointestinal disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT01794793/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT01794793/SAP_001.pdf
  • Informed Consent Form (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT01794793/ICF_002.pdf